CLINICAL TRIAL: NCT00184379
Title: Effects of Psychoeducation of Relatives to Patients With Serious Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4.2005.389
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Mental Disorder; Depressive Disorder; Schizophrenia
Keywords: Family; Coping Skills; Psychoeducation; Stress, Psychological; Health Education
MeSH Terms: conditions — Mental Disorders; Depressive Disorder; Schizophrenia; Stress, Psychological; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1 S+E (Experimental): Relatives of patients with schizophrenia, who receive education
  Interventions: Behavioral: Psychoeducation
- 2 S-E (No Intervention): Relatives of patients with schizophrenia, who do not receive education
- 3 B+E (Experimental): Relatives of patients with bipolar disorder, who receive education
  Interventions: Behavioral: Psychoeducation
- 4 B-E (No Intervention): Relatives of patients with bipolar disorder, who do not receive education

INTERVENTIONS:
Behavioral: Psychoeducation — Structured disorder-related educational program for relatives
  Arms: 1 S+E; 3 B+E

SUMMARY:
The purpose of this study is to determine the effects of psychoeducation for relatives to patients with serious mental illness.

DETAILED DESCRIPTION:
The main aim of the study is to compare the effects of group psychoeducation for relatives to patients with serious mental illness with a waiting list control group. The main hypothesis is whether psychoeducation in groups has effects on the stress experience and coping style in the relatives. The relatives will receive group education in 6 weekly sessions. We will measure stress experience, coping style and the relatives' health condition before the sessions, after the sessions and at one year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Relatives to patients having a psychotic or bipolar disorder
* Good Norwegian language skills
* Consent to participate
* The patients' consent for their relatives to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
ECI (Experience of Caregiving Inventory) (Smuckler et al,1994) | 0-6 months
COOP/WONCA (Bowling, 1995) | 0-6 months
Selection of questions from COPE (Carver et al. 1989) | 0-6 months
Evaluation-questions | 0-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Olav M Linaker, MD Prof, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Østmarka Psychiatric Department, St. Olavs Hospital, University Hospital of Trondheim, Trondheim, Norway

REFERENCES:
- [Result] Moller T, Gudde CB, Folden GE, Linaker OM. The experience of caring in relatives to patients with serious mental illness: gender differences, health and functioning. Scand J Caring Sci. 2009 Mar;23(1):153-60. doi: 10.1111/j.1471-6712.2008.00605.x. Epub 2009 Jan 21. PMID 19192243